CLINICAL TRIAL: NCT00597779
Title: Extramedullary vs. Intramedullary Devices in the Treatment of Unstable Intertrochanteric Hip Fractures
Brief Title: Randomized Comparison of 2 Fixation Techniques for Unstable Intertrochanteric Hip Fractures
Acronym: EMvsIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rudy Reindl (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor-Investigator, Rudy Reindl, MD FRCSC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN #07-065
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Hip Fractures
Keywords: intertrochanteric fractures
MeSH Terms: conditions — Hip Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EM device (Active Comparator): Extramedullary Device (EM)
  Interventions: Device: Dynamic Hip Screw (DHS); Trochanteric Fixation Nail (TFN)
- IM device (Active Comparator): Intramedullary Device (IM)
  Interventions: Device: Dynamic Hip Screw (DHS); Trochanteric Fixation Nail (TFN)

INTERVENTIONS:
Device: Dynamic Hip Screw (DHS); Trochanteric Fixation Nail (TFN) — Surgical stabilization of unstable intertrochanteric hip fractures using two commonly used implant categories
  Other Names: Extramedullary plate/ screw device , Intramedullary nail

SUMMARY:
The purpose of this study is to compare the clinical and radiological outcome of patients that are treated with two different orthopedic implants. The study population will consist of patients that have sustained unstable hip fractures. The two different implants will be randomly assigned.

The null hypothesis states that there should not be any significant differences between the two implants.

DETAILED DESCRIPTION:
Intertrochanteric hip fractures are common injuries in the elderly population. They often signify generalized physical deterioration. Operative management has become the standard of care to prevent life threatening complications and dates back to the 1940's. The design of implants has evolved significantly since then.

The sliding hip screw replaced static fixation of the femoral head in the 1950's. As a result of this improvement in design, failures have been reduced to 9-16%. The sliding hip screw allows for stable collapse of the femoral neck. This can lead to significant shortening of the proximal femur in comminuted fractures.

Current treatment modalities focus on obtaining a satisfactory union of the fracture, often at the expense of anatomical alignment. Severely comminuted fractures treated with a standard plate-hip-screw device thus commonly result in significant degrees of mal-union and shortening. In the past, implants designed to restore and maintain the anatomy of the hip have resulted in high failure rates with the implant breaking out of the femoral head. In the mid 1980's, recognition of this led to the development of various intramedullary devices for fixation of these fractures. The weight-bearing portion of the implant is therefore shifted medially, resulting in reduced lever forces on the implant and femur. Additionally, the IM device does not rely on fixation to the lateral cortex of the femur with screws. From a biomechanical standpoint, the intramedullary device has distinct advantages, as it is a load- sharing device more closely located to the axis of weight bearing than the plate-hip-screw device.

Advances in intramedullary designs have been promising, but the clinical results variable. The relatively high rate of fracture at the tip, specifically at the level of the locking bolts, has hampered the widespread popularity of intramedullary devices. Additionally, the large diameter of the proximal aspect of the implants required extensive reaming of the greater trochanter and partial detachment of the gluteus medius. This may lead to abductor weakness and a Trendelenburg gait. Some studies have found increased re-operation rates for these early hip-nail devices compared to the plate -hip-screw implant. Other studies have shown decreased blood loss and operative time with the nails. A meta-analysis of the literature favors the sliding hip screw design. Unfortunately, most studies focus on radiological failure rate rather than patient function and relate to the first generation of IM devices.

The newest generation of nails (like the IM studied here) has attempted to correct the shortcomings of earlier designs. The proximal aspect of the nail diameter is minimized. The distal locking screw is located far away from the distal end of the nail and the locking bolt is placed in an oblique fashion. Design alterations to the femoral head fixation portion of the nail by using a helical blade rather than a screw may improve fixation in the femoral head. These new designs seem to compare favorably in recent clinical tests. Early mobilization for patients with the intramedullary device (IM) seems to be better.

Results of the pilot study indicate an earlier return to full mobility and shorter operating time in the IM group. This study included all intertrochanteric fracture types and did not demonstrate a clear benefit of the IM in many other parameters. The currently proposed multi-centre study will focus on the unstable A2 intertrochanteric fracture pattern.

Considering the significantly increased cost of the new intramedullary devices compared to the standard plate-hip-screw, a significant overall improvement in patient function should be realized before the general use of these new devices could be recommended.

ELIGIBILITY:
Inclusion Criteria:

1. 55 years or older
2. Type A2 Intertrochanteric fractures
3. Mono trauma
4. Medically fit for surgery
5. Less than 2 weeks post fracture

Exclusion Criteria:

1. Fractures due to malignancy
2. Non-ambulatory pre-fracture
3. Severe dementia
4. Limited life expectancy due to significant medical co-morbidities
5. Medical contraindication to surgery
6. Inability to comply with rehabilitation of form completion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Timed 2 minute walking distance | 6 weeks, 3 months, 6 months and 12 months
TUG (Time up and go) test | 6 weeks, 3 months, 6 months and 12 months
Trendelenburg's test: pelvic drop | 6 weeks, 3 months, 6 months and 12 months
Fracture classification: Mueller/ AO, displacement, time to union, heterotopic ossification and shortening. | 6 weeks, 3 months, 6 months and 12 months
FIM (Functional Independence Measure) | 6weks, 3months, 6months and 12months
LEM (Lower Extremity Measure) | 6weeks, 3months, 6months and 12 months

SECONDARY OUTCOMES:
Secondary Outcome Variable: Transfusions | 6 weeks, 3 months, 6 months and 12 months
Pre and Post operative Hgb | 6 weeks, 3 months, 6 months and 12 months
Complications/ Re-operation | 6 weeks, 3 months, 6 months and 12 months
Length of surgery and hospital stay | 6 weeks, 3 months, 6 months and 12 months
Weight bearing status post-op | 6 weeks, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Reindl, MD FRCSC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre - Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Reindl R, Harvey EJ, Berry GK, Rahme E; Canadian Orthopaedic Trauma Society (COTS). Intramedullary Versus Extramedullary Fixation for Unstable Intertrochanteric Fractures: A Prospective Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Dec 2;97(23):1905-12. doi: 10.2106/JBJS.N.01007. PMID 26631990